CLINICAL TRIAL: NCT02311439
Title: Induction Chemotherapy, Fluorouracil, Leucovorin, Oxaliplatin and Irinotecan (FOLFIRINOX) Followed With Concurrent Capecitabine and Radiation Therapy in Treatment of Patients With Inoperable Locally Advanced Cancer Pancreas
Brief Title: Induction Chemotherapy, FOLFIRINOX Followed With Concurrent Capecitabine and Radiation Therapy in Inoperable Locally Advanced Cancer of the Pancreas
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Allam Abdelhamed Mohamed, Dr, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAP001
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Cancer of Pancreas
Keywords: Locally advanced pancreatic cancer; Chemotherapy; Radiotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — folfirinox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FOLFIRINOX + CRT (Experimental): FOLFIRINOX regimen, consisted of oxaliplatin, irinotecan, leucovorin and fluorouracil (5-FU), for 4 cycles, followed by consolidation radiotherapy concurrent with capecitabine 625mg/m2 BID in non-progressed cases, in treating patients with locally advanced cancer pancreas.
  Interventions: Drug: FOLFIRINOX + CRT

INTERVENTIONS:
Drug: FOLFIRINOX + CRT — Induction 4 times chemotherapy, FOLFIRINOX regimen, consisted of Oxaliplatin at a dose of 85 mg/m2 D1, 2-hour I.V + Irinotecan 180 mg/m2 D1 90-minute I.V. + Leucovorin 200 mg/m2 2- hour I.V, D1,2 + (5-FU) dosed at 400 mg/m2, administered as an intravenous bolus on day 1 and day 2, followed by a continuous intravenous infusion of 600 /m2 over a 20- hours period on day 1 and day 2. Treatment will be administered every 2 weeks. G-CSF will be administrated according to the need.
  In non-progressed cases, will be followed by consolidation concurrent radiotherapy with capecitabine 625 mg/m2 BID.
  Radiotherapy :
  A fractionated dose of 50.4Gy /28 fractions/15 MeV photon energy generated by Dual-energetic Linear Accelerator.

SUMMARY:
This prospective cohort, phase II, trial is studying induction chemotherapy combination, FOLFIRINOX regimen, consisted of oxaliplatin, irinotecan, leucovorin and fluorouracil (5-FU), for 4 cycles, followed by consolidation concurrent radiotherapy with capecitabine in non-progressed cases, in treating patients with locally advanced cancer pancreas.

DETAILED DESCRIPTION:
Design & Methodology:

1. Nature of the study:

   It is ( prospective cohort study).
2. Study subjects:

   *Target Population: Patients, fulfilling the inclusion criteria for the research, will be selected from Assiut clinical oncology department in Assiut University Hospitals.
   * Sample size:

     20 patients.
   * Characteristics of subjects:

     * Inclusion criteria:

   Disease characteristics:
   * Histological and radiological confirmation of locally advanced cancer pancreas
   * Inoperable disease
   * Disease must be able to be encompassed within a radical radiotherapy treatment volume
   * Not metastatic

   Patient characteristics:
   * ECOG performance status 0 or 1
   * Life expectancy > 3 months.
   * Glomerular filtration rate ≥ 60 mL/min.
   * WBC > 3,000/mm³.
   * Absolute neutrophil count > 1,500/mm³.
   * Hemoglobin > 10.0 g/dL.
   * Platelet count > 100,000/mm³.
   * Alkaline phosphatase ≤ 1.5 times upper limit of normal (ULN)
   * Gamma-glutamyl-transferase < 1.5 times ULN.
   * Transaminases ≤ 1.5 times ULN.
   * Bilirubin ≤ 1.5 times ULN.
   * No medically unstable conditions (e.g., unstable diabetes, uncontrolled arterial hypertension, infection, hypercalcemia, or ischemic heart disease)
   * Not pregnant or nursing.
   * No other previous or current malignant disease likely to interfere with protocol treatment or comparisons
   * No prior chemotherapy or radiotherapy.
3. Patients & Methods:

   Patients are randomized to one treatment arm. Induction 4 times chemotherapy, FOLFIRINOX regimen, consisted of Oxaliplatin at a dose of 85 mg/m2 on day 1 only, administered as a 2-hour intravenous infusion, with the addition, after 30 minutes, of Irinotecan at a dose of 180 mg/m2 on day 1 only given as a 90-minute intravenous infusion. immediately will be followed by Leucovorin at a dose of 200 mg/m2, given as a 2- hour intravenous infusion, day 1 and day 2 This treatment will be followed by fluorouracil (5-FU) dosed at 400 mg/m2, administered as an intravenous bolus on day 1 and day 2, followed by a continuous intravenous infusion of 600 /m2 over a 20- hours period on day 1 and day 2. Treatment will be administered every 2 weeks. G-CSF will be administrated according to the need.

   In non-progressed cases, induction chemotherapy will be followed by consolidation radiotherapy concurrent with capecitabine 625 mg/m2 BID.

   Radiotherapy :

   A fractionated dose of 50.4Gy /28 fraction/15 MeV photon energy generated by Dual-energetic Linear Accelerator.
   * Gross Target Volume (GTV): visible tumor and lymph nodes.
   * Clinical Target Volume (CTV): [tumor/ affected lymph node + 1-2 cm] + regional lymphatics Lymphatics :corpus: upper and lower pancreaticoduodenal, superior and inferior pancreatic, celiac Head: corpus lymphatics + porta hepatis lymphatics Tail: corpus lymphatics (except pancreaticoduodenal LN) + splenic hilum LN
   * PTV: CTV + 1-1.5 cm

     * All patients will undergo a complete classical evaluation at the time of presentation which will be enrolled in a separate sheet for each patient. This will include a detailed history with estimation of the age of onset, the duration of the disease,.
     * Detailed physical examination will be carried out Treatment evaluation . Laboratory examination include
     * complete blood count (CBC),
     * liver function test (LFT)
     * Renal function test (RFT),
     * Serum electrolytes at presentation and before each cycle of chemotherapy.

   Radiographic examination include
   * Abdominal Multi Detector Computed Tomography (MDCT Abdomen )
   * Chest X-ray Before starting treatment, 2 weeks after ending phase 1 of treatment then 4 weeks after ending phase 2 of treatment then every 3 months for 18 months.

     ● Bone scan will be done in those complaining from bone pain; elevated serum alkaline phosphatase or transaminase level
   * Quality of life is assessed at baseline, monthly for 6 months, and then at each follow-up visit.

   After completion of study treatment, patients are followed periodically. Response Assessment : will be carried out, using (RECIST) Response Evaluation Criteria In Solid Tumors, Version 1.1 Chemotherapy Toxicity Assessment: will be carried out, using (CTCAE) Common Terminology Criteria for Adverse Events, Version 4.0
4. Data analysis:

Data will be analysed using the computer program, Statistical Package for the Social Science (SPSS V.16).

Expected outcomes:

The outcome of the study will be compared statistically with previous local and international trails.

Ethical considerations:

1. Risk-benefit assessment:

   There is an acceptable risk may affect the patient in this research study as regard the acceptable side effects of Gemcitabine, Oxaliplatin and radiotherapy.
2. Confidentiality:

   Any data taken from the patient either from history, the examination or the investigations will be very confidential.
3. Research statement:

   All patients subjected to this study will be informed about the procedures of the research.
4. Informed consent:

   The study procedures will be discussed to all patients and consent will be taken from them.
5. Other ethical concerns:

The research will be conducted only by scientifically qualified and trained personnel.

ELIGIBILITY:
Inclusion Criteria:

* Disease characteristics:

  * Histological and radiological confirmation of locally advanced cancer pancreas
  * Inoperable disease
  * Disease must be able to be encompassed within a radical radiotherapy treatment volume
  * Not metastatic

Patient characteristics:

* ECOG performance status 0 or 1
* Life expectancy > 3 months.
* Glomerular filtration rate ≥ 60 mL/min.
* WBC > 3,000/mm³.
* Absolute neutrophil count > 1,500/mm³.
* Hemoglobin > 10.0 g/dL.
* Platelet count > 100,000/mm³.
* Alkaline phosphatase ≤ 1.5 times upper limit of normal (ULN)
* Gamma-glutamyl-transferase < 1.5 times ULN.
* Transaminases ≤ 1.5 times ULN.
* Bilirubin ≤ 1.5 times ULN.
* No medically unstable conditions (e.g., unstable diabetes, uncontrolled arterial hypertension, infection, hypercalcemia, or ischemic heart disease)
* Not pregnant or nursing.
* No other previous or current malignant disease likely to interfere with protocol treatment or comparisons
* No prior chemotherapy or radiotherapy.

Exclusion Criteria:

* ECOG performance status > 2
* Life expectancy < 3 months.
* Glomerular filtration rate < 30 mL/min.
* Absolute neutrophil count < 1,500/mm³.
* Alkaline phosphatase > 1.5 times upper limit of normal (ULN)
* Gamma-glutamyl-transferase > 1.5 times ULN.
* Transaminases>1.5 times ULN.
* Bilirubin >1.5 times ULN.
* medically unstable conditions (e.g., unstable diabetes, uncontrolled arterial hypertension, infection, hypercalcemia, or ischemic heart disease)
* pregnant or nursing.
* prior chemotherapy or radiotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-11 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability of FOLFIRINOX plus Concurrent Radiotherapy with Capecitabine | 6 months after enrolment
  will be carried out, using (CTCAE) Common Terminology Criteria for Adverse Events, Version 4.0

SECONDARY OUTCOMES:
Tumor response | 6 months after enrolment
  will be carried out, using (RECIST) Response Evaluation Criteria In Solid Tumors, Version 1.1

OTHER OUTCOMES:
Progression Free Survival | 6 months after finishing protocol
Number of Cases will have radical surgery | 6 months after enrolment

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospitals, Asyut, Asyut Governorate, Egypt